CLINICAL TRIAL: NCT02955797
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Toddlers 12 to 23 Months of Age.
Brief Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine in Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET51; U1111-1161-2935 (Other: WHO); 2016-000749-30 (EudraCT Number)
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; MenACYW Conjugate vaccine; Nimenrix®; Menjugate®
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal vaccine naive toddlers aged 12 to 23 months received a single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Group 2 (Meningococcal Vaccine-Naive): Nimenrix® (Experimental): Healthy, meningococcal vaccine naive toddlers aged 12 to 23 months received a single dose of Nimenrix® vaccine on Day 0.
  Interventions: Biological: Meningococcal polysaccharide groups A, C, W-135 and Y Conjugate vaccine
- Group 3 (MenC-Primed): MenACYW Conjugate Vaccine (Experimental): Healthy, meningococcal C vaccine primed toddlers aged 12 to 23 months received a single dose of MenACYW Conjugate vaccine on Day 0.
  Interventions: Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine
- Group 4 (MenC-Primed): Nimenrix® (Experimental): Healthy, meningococcal C vaccine primed toddlers aged 12 to 23 months received a single dose of Nimenrix® vaccine on Day 0.
  Interventions: Biological: Meningococcal polysaccharide groups A, C, W-135 and Y Conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — 0.5 milliliter (mL), Intramuscular
  Other Names: MenACYW Conjugate vaccine
  Arms: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine
Biological: Meningococcal polysaccharide groups A, C, W-135 and Y Conjugate vaccine — 0.5 mL, Intramuscular
  Other Names: Nimenrix®
  Arms: Group 2 (Meningococcal Vaccine-Naive): Nimenrix®
Biological: Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid Conjugate Vaccine — 0.5 mL, Intramuscular
  Other Names: MenACYW Conjugate vaccine
  Arms: Group 3 (MenC-Primed): MenACYW Conjugate Vaccine
Biological: Meningococcal polysaccharide groups A, C, W-135 and Y Conjugate vaccine — 0.5 mL, Intramuscular
  Other Names: Nimenrix®
  Arms: Group 4 (MenC-Primed): Nimenrix®

SUMMARY:
The purpose of the study was to evaluate the immunogenicity and describe the safety of a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine compared to the licensed Meningococcal polysaccharide groups A, C, W-135 and Y (Nimenrix®) Conjugate vaccine in toddlers 12 to 23 months of age in the European Union (EU). The toddlers were either meningococcal vaccine naïve or had received monovalent meningococcal C (MenC) vaccination during infancy to evaluate any potential impact of the meningococcal vaccine background on the immunogenicity and safety profile of the investigational product.

Primary Objectives:

* To demonstrate the non-inferiority of the antibody response to meningococcal serogroups A, C, Y, and W after a single dose of MenACYW Conjugate vaccine or Nimenrix® in toddlers who either were meningococcal vaccine naïve or had received monovalent MenC vaccination during infancy.
* To demonstrate the non-inferiority of the antibody response to meningococcal serogroups A, C, Y, and W after a single dose of MenACYW Conjugate vaccine or Nimenrix® in meningococcal vaccine naïve toddlers.

Secondary Objectives:

* To compare the antibody responses (geometric mean titers [GMTs]) to meningococcal serogroups A, C, Y, and W after a dose of MenACYW Conjugate vaccine or Nimenrix® as measured by serum bactericidal assay using human complement (hSBA) in toddlers who either were meningococcal vaccine naïve or had received monovalent MenC vaccination during infancy.
* To compare the antibody responses (GMTs) to meningococcal serogroups A, C, Y, and W after a dose of MenACYW Conjugate vaccine or Nimenrix® as measured by hSBA in meningococcal vaccine naïve toddlers.
* To compare the antibody responses (GMTs) to meningococcal serogroups A, C, Y, and W after a dose of MenACYW Conjugate vaccine or Nimenrix® as measured by hSBA in toddlers who received monovalent MenC vaccination during infancy.

DETAILED DESCRIPTION:
Healthy toddlers were randomized depending on their meningococcal priming vaccination background (either meningococcal vaccine naïve or primed with MenC) and received a single dose of either MenACYW Conjugate vaccine or Nimenrix®. They were assessed for immunogenicity at baseline (pre-vaccination) and 30 to 44 days post-vaccination. Safety information were collected post-vaccination and throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 to 23 months on the day of the first study visit.
* Participants had received all recommended standard-of-care non-meningococcal vaccinations according to his/her age as per local regulations.
* Informed consent form (ICF) had been signed and dated by the parent/legally acceptable representative.
* Participant and parent/legally acceptable representative were able to attend all scheduled visits and complied with all trial procedures.
* Covered by health insurance if required by local regulations.
* Participants had received any meningococcal vaccine in the second year of life (i.e., from 12 months of age).
* For Inclusion in Groups 1 and 2: Participants must not had received any vaccination against meningococcal disease with either a trial vaccine or a licensed meningococcal vaccine (i.e., polyvalent, polysaccharide, or Conjugate meningococcal vaccine containing serogroups A, C, W, Y, B; or any monovalent or bivalent meningococcal vaccine).
* For Inclusion in Groups 3 and 4: Participants must had previously received at least 1 dose of licensed monovalent meningococcal C Conjugate (MenC) vaccine during infancy (i.e., before 12 months of age).

Exclusion Criteria:

* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which may be received at least 2 weeks before or after study investigational vaccines. This exception included monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* For Groups 1 and 2 only: Vaccination against meningococcal disease with either a trial vaccine or a licensed meningococcal vaccine (i.e., polyvalent, polysaccharide, or Conjugate meningococcal vaccine containing serogroups A, C, W, Y, B; or any monovalent or bivalent meningococcal vaccine).
* For Groups 3 and 4 only: Vaccination against meningococcal disease with either a trial vaccine or a licensed meningococcal vaccine (i.e., polyvalent, polysaccharide, or Conjugate meningococcal vaccine containing serogroups A, C, W, Y, B; or any monovalent B meningococcal vaccine), except licensed monovalent meningococcal C Conjugate (MenC) vaccination received during infancy.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants travelling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine.
* Personal history of Guillain-Barré Syndrome.
* Verbal report of thrombocytopenia, as reported by the parent/legally acceptable representative contraindicating intramuscular vaccination in the Investigator's opinion.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw - Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 918 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (33):
- Finland (10):
  - Investigational Site 309, Espoo
  - Investigational Site 301, Helsinki
  - Investigational Site 306, Helsinki
  - Investigational Site 302, Jarvenpaa
  - Investigational Site 304, Kokkola
  - Investigational Site 307, Oulu
  - Investigational Site 303, Pori
  - Investigational Site 305, Seinäjoki
  - Investigational Site 308, Tampere
  - Investigational Site 310, Turku
- Germany (12):
  - Investigator Site 412, Aschaffenburg
  - Investigator Site 411, Bönnigheim
  - Investigator Site 401, Bramsche
  - Investigator Site 407, Bretten
  - Investigator Site 413, Datteln
  - Investigator Site 408, Goch
  - Investigator Site 406, Hamburg
  - Investigator Site 415, Hamburg
  - Investigator Site 404, Ludwigsfelde
  - Investigator Site 409, Rosenheim
  - Investigator Site 402, Tauberbischofsheim
  - Investigator Site 403, Tauberbischofsheim
- Hungary (6):
  - Investigational Site 102, Budapest
  - Investigational Site 101, Budapest
  - Investigational Site 104, Győr
  - Investigational Site 105, Miskolc
  - Investigational Site 103, Szeged
  - Investigational Site 106, Székesfehérvár
- Spain (5):
  - Investigator Site 203, Barcelona
  - Investigator Site 204, Galicia
  - Investigator Site 205, Madrid
  - Investigator Site 202, Madrid
  - Investigator Site 201, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 34 centers in Spain, Hungary, Germany and Finland from 24 February 2017 to 21 September 2017.
Pre-assignment Details: A total of 918 participants were enrolled and randomized in the study.
Groups:
- Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine: Healthy, meningococcal vaccine naive toddlers aged 12 to 23 months received a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y and W) Tetanus Toxoid (MenACYW) Conjugate vaccine on Day 0.
- Group 2 (Meningococcal Vaccine-Naive): Nimenrix®: Healthy, meningococcal vaccine naive toddlers aged 12 to 23 months received a single dose of Meningococcal polysaccharide groups A, C, W-135 and Y (Nimenrix®) Conjugate vaccine on Day 0.
- Group 3 (MenC-Primed) MenACYW Conjugate Vaccine: Healthy, meningococcal C (MenC) vaccine primed toddlers aged 12 to 23 months received a single dose of MenACYW Conjugate vaccine on Day 0.
Period: Overall Study
Arm/Group | Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine | Group 2 (Meningococcal Vaccine-Naive): Nimenrix® | Group 3 (MenC-Primed) MenACYW Conjugate Vaccine | Group 4 (MenC-Primed): Nimenrix®
Started | 306 | 306 | 203 | 103
Safety Analysis Set (SafAS) (SafAS:participants who received at least 1 dose of study vaccine(s) & had any safety data available.) | 303 | 306 | 203 | 102
Per Protocol Analysis Set (PPAS) (Who had at least 1 dose of vaccine, valid post-vaccination serology data with no protocol deviation.) | 293 | 296 | 198 | 99
Completed | 303 | 303 | 203 | 101
Not Completed | 3 | 3 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine | Group 2 (Meningococcal Vaccine-Naive): Nimenrix® | Group 3 (MenC-Primed): MenACYW Conjugate Vaccine | Group 4 (MenC-Primed): Nimenrix® | Total
Number analyzed (Participants) | 306 | 306 | 203 | 103 | 918
Age, Continuous [Mean (Standard Deviation); unit: months] | 16.1 (3.32) | 16.2 (3.19) | 14.0 (3.01) | 13.8 (2.72) | 15.4 (3.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 145 | 97 | 53 | 435
  Male | 166 | 161 | 106 | 50 | 483
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 1 | 3
  White | 115 | 132 | 197 | 99 | 543
  More than one race | 2 | 3 | 5 | 2 | 12
  Unknown or Not Reported | 188 | 168 | 0 | 0 | 356
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 0 | 0 | 95 | 50 | 145
  Finland | 188 | 168 | 0 | 0 | 356
  Germany | 118 | 138 | 0 | 0 | 256
  Spain | 0 | 0 | 108 | 53 | 161

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Antibody Titers Greater Than or Equal to (>=) 1:8 Against Meningococcal Serogroups A, C, Y, and W in Toddlers Who Either Were Meningococcal Vaccine Naïve or Had Received Monovalent MenC Vaccination During Infancy
Description: Antibody titers against Meningococcal Serogroups A, C, Y, and W were measured by serum bactericidal assay using human complement (hSBA). Data for this outcome measure were planned to be analyzed for the pooled population of MenACYW Conjugate vaccine and Nimenrix® reporting groups.
Time Frame: Day 30 (post-vaccination)
Population: Per-protocol analysis set (PPAS) defined for accessing ACYW immune response data for participants who received at least one dose of study vaccine and had a valid post-vaccination serology result. Participants with pre-defined protocol deviations were excluded. Here, "Number analyzed" = participants with available data for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- MenACYW Conjugate Vaccine (Groups 1 and 3): All healthy meningococcal-vaccine naive and meningococcal C vaccine primed toddlers aged 12 to 23 months who received a single dose of MenACYW Conjugate vaccine on Day 0.
- Nimenrix® (Groups 2 and 4): All meningococcal-vaccine naive and meningococcal C vaccine primed participants who a single dose of Nimenrix® vaccine on Day 0.
Arm/Group | MenACYW Conjugate Vaccine (Groups 1 and 3) | Nimenrix® (Groups 2 and 4)
Number analyzed (Participants) | 491 | 395
percentage of participants
  Serogroup A: number analyzed (Participants) | 490 | 394
  Serogroup A | 90.4 [87.4 to 92.9] | 91.6 [88.4 to 94.2]
  Serogroup C: number analyzed (Participants) | 489 | 394
  Serogroup C | 99.2 [97.9 to 99.8] | 85.5 [81.7 to 88.9]
  Serogroup Y: number analyzed (Participants) | 490 | 395
  Serogroup Y | 94.3 [91.8 to 96.2] | 91.6 [88.5 to 94.2]
  Serogroup W: number analyzed (Participants) | 489 | 394
  Serogroup W | 84.9 [81.4 to 87.9] | 84.0 [80.0 to 87.5]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine (Groups 1 and 3) vs Nimenrix® (Groups 2 and 4); Serogroup A; Test type: Non-Inferiority — 95% confidence interval (CI) was stratified on the priming status (meningococcal vaccine naïve or primed monovalent MenC vaccination during infancy) and calculated using the Wald method (normal approximation). Weighted average of the difference over strata was calculated using the Minimal Risk weights with the null variance method. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference between the 2 percentages was greater than (>) -10%; Percentage difference = -2.03, 95% CI 2-sided [-5.84 to 1.78]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine (Groups 1 and 3) vs Nimenrix® (Groups 2 and 4); Serogroup C; Test type: Non-Inferiority — 95% CI was stratified on the priming status (meningococcal vaccine naïve or primed monovalent MenC vaccination during infancy) and calculated using the Wald method (normal approximation). Weighted average of the difference over strata was calculated using the Minimal Risk weights with the null variance method. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference between the 2 percentages was > -10%; Percentage difference = 12.1, 95% CI 2-sided [8.16 to 16.1]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine (Groups 1 and 3) vs Nimenrix® (Groups 2 and 4); Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage difference = 2.42, 95% CI 2-sided [-1.34 to 6.19]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine (Groups 1 and 3) vs Nimenrix® (Groups 2 and 4); Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Percentage difference = 0.458, 95% CI 2-sided [-4.37 to 5.28]

2. Primary Outcome: Percentage of Participants With Antibody Titers >=1:8 Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® in Meningococcal Vaccine Naïve Toddlers
Description: Antibody titers against Meningococcal Serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here, "Number analyzed" = participants with available data for each specified category. Data for this outcome measure were not planned to be collected and analyzed for MenC-primed reporting groups (Groups 3 and 4).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine | Group 2 (Meningococcal Vaccine-Naive): Nimenrix®
Number analyzed (Participants) | 293 | 296
percentage of participants
  Serogroup A: number analyzed (Participants) | 293 | 295
  Serogroup A | 90.8 [86.9 to 93.8] | 89.5 [85.4 to 92.7]
  Serogroup C: number analyzed (Participants) | 293 | 295
  Serogroup C | 99.3 [97.6 to 99.9] | 81.4 [76.4 to 85.6]
  Serogroup Y | 93.2 [89.7 to 95.8] | 91.6 [87.8 to 94.5]
  Serogroup W | 83.6 [78.9 to 87.7] | 83.4 [78.7 to 87.5]
Statistical Analysis 1: Comparison: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine vs Group 2 (Meningococcal Vaccine-Naive): Nimenrix®; Serogroup A; Test type: Non-Inferiority — 95% CI of the difference in percentages was computed using the Wilson Score method without continuity correction. Non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI of the difference between the 2 percentages was > -10%; Percentage difference = 1.3, 95% CI 2-sided [-3.6 to 6.2]
Statistical Analysis 2: Comparison: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine vs Group 2 (Meningococcal Vaccine-Naive): Nimenrix®; Serogroup C; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage difference = 18, 95% CI 2-sided [13.6 to 22.8]
Statistical Analysis 3: Comparison: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine vs Group 2 (Meningococcal Vaccine-Naive): Nimenrix®; Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage difference = 1.6, 95% CI 2-sided [-2.76 to 6.03]
Statistical Analysis 4: Comparison: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine vs Group 2 (Meningococcal Vaccine-Naive): Nimenrix®; Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage difference = 0.2, 95% CI 2-sided [-5.85 to 6.18]

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W in Toddlers Who Either Were Meningococcal Vaccine Naïve or Had Received Monovalent MenC Vaccination During Infancy
Description: Antibody titers against Meningococcal Serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here, "Number analyzed" = participants with available data for each specified category. Data for this outcome measure were planned to be analyzed for the pooled population of MenACYW Conjugate vaccine and Nimenrix® reporting groups.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- Nimenrix® (Groups 2 and 4): All meningococcal vaccine naive and meningococcal C vaccine primed participants who a single dose of Nimenrix® vaccine on Day 0.
Arm/Group | MenACYW Conjugate Vaccine (Groups 1 and 3) | Nimenrix® (Groups 2 and 4)
Number analyzed (Participants) | 491 | 395
titers (1/dilution)
  Serogroup A: number analyzed (Participants) | 490 | 394
  Serogroup A | 29.9 [26.9 to 33.2] | 34.5 [30.5 to 39.0]
  Serogroup C: number analyzed (Participants) | 489 | 394
  Serogroup C | 880 [748 to 1035] | 77.1 [60.7 to 98.0]
  Serogroup Y: number analyzed (Participants) | 490 | 395
  Serogroup Y | 41.7 [37.5 to 46.5] | 31.9 [28.4 to 36.0]
  Serogroup W: number analyzed (Participants) | 489 | 394
  Serogroup W | 24.4 [21.8 to 27.5] | 17.7 [15.8 to 19.8]
Statistical Analysis 1: Comparison: MenACYW Conjugate Vaccine (Groups 1 and 3) vs Nimenrix® (Groups 2 and 4); Serogroup A; Test type: Other — 95% CI of the ratio of post-vaccination GMTs was stratified on the priming vaccination status (meningococcal vaccine naïve or primed monovalent MenC vaccination) and calculated using an analysis of variance (ANOVA) model of log10-transformed titers; GMT Ratio = 0.819, 95% CI 2-sided [0.697 to 0.963]
Statistical Analysis 2: Comparison: MenACYW Conjugate Vaccine (Groups 1 and 3) vs Nimenrix® (Groups 2 and 4); Serogroup C; Test type: Other — 95% CI of the ratio of post-vaccination GMTs was stratified on the priming vaccination status (meningococcal vaccine naïve or primed monovalent MenC vaccination) and calculated using an ANOVA model of log10-transformed titers; GMT Ratio = 7.59, 95% CI 2-sided [6.05 to 9.52]
Statistical Analysis 3: Comparison: MenACYW Conjugate Vaccine (Groups 1 and 3) vs Nimenrix® (Groups 2 and 4); Serogroup Y; Test type: Other — [test comment as in outcome 3, analysis 2]; GMT Ratio = 1.28, 95% CI 2-sided [1.09 to 1.51]
Statistical Analysis 4: Comparison: MenACYW Conjugate Vaccine (Groups 1 and 3) vs Nimenrix® (Groups 2 and 4); Serogroup W; Test type: Other — [test comment as in outcome 3, analysis 2]; GMT Ratio = 1.32, 95% CI 2-sided [1.12 to 1.56]

4. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® in Vaccine Naive Toddlers
Description: Antibody titers against Meningococcal Serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here, "Number analyzed" = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine | Group 2 (Meningococcal Vaccine-Naive): Nimenrix®
Number analyzed (Participants) | 293 | 296
titers (1/dilution)
  Serogroup A: number analyzed (Participants) | 293 | 295
  Serogroup A | 28.7 [25.2 to 32.6] | 28.0 [24.4 to 32.1]
  Serogroup C: number analyzed (Participants) | 293 | 295
  Serogroup C | 436 [380 to 500] | 26.4 [22.5 to 31.0]
  Serogroup Y | 38.0 [33.0 to 43.9] | 32.2 [28.0 to 37.0]
  Serogroup W | 22.0 [18.9 to 25.5] | 16.4 [14.4 to 18.6]
Statistical Analysis 1: Comparison: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine vs Group 2 (Meningococcal Vaccine-Naive): Nimenrix®; Serogroup A; Test type: Other; GMT Ratio = 1.03, 95% CI 2-sided [0.85 to 1.24]
Statistical Analysis 2: Comparison: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine vs Group 2 (Meningococcal Vaccine-Naive): Nimenrix®; Serogroup C; Test type: Other; GMT Ratio = 16.5, 95% CI 2-sided [13.4 to 20.4]
Statistical Analysis 3: Comparison: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine vs Group 2 (Meningococcal Vaccine-Naive): Nimenrix®; Serogroup Y; Test type: Other; GMT Ratio = 1.18, 95% CI 2-sided [0.97 to 1.44]
Statistical Analysis 4: Comparison: Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine vs Group 2 (Meningococcal Vaccine-Naive): Nimenrix®; Serogroup W; Test type: Other; GMT Ratio = 1.34, 95% CI 2-sided [1.1 to 1.63]

5. Secondary Outcome: Geometric Mean Titers of Antibodies Against Meningococcal Serogroups A, C, Y, and W Following Vaccination With MenACYW Conjugate Vaccine or Nimenrix® in Toddlers Who Had Received Monovalent MenC Vaccination During Infancy
Description: Antibody titers against Meningococcal Serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 30 (post-vaccination)
Population: Analysis was performed on PPAS. Here, "Number analyzed" = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 3 (MenC-Primed): MenACYW Conjugate Vaccine | Group 4 (MenC-Primed): Nimenrix®
Number analyzed (Participants) | 198 | 99
titers (1/dilution)
  Serogroup A: number analyzed (Participants) | 197 | 99
  Serogroup A | 31.8 [26.5 to 38.1] | 64.0 [50.9 to 80.5]
  Serogroup C: number analyzed (Participants) | 196 | 99
  Serogroup C | 2514 [1875 to 3372] | 1883 [1276 to 2779]
  Serogroup Y: number analyzed (Participants) | 197 | 99
  Serogroup Y | 48.0 [40.6 to 56.7] | 31.3 [24.8 to 39.5]
  Serogroup W: number analyzed (Participants) | 196 | 98
  Serogroup W | 28.7 [23.8 to 34.5] | 22.3 [17.7 to 28.2]
Statistical Analysis 1: Comparison: Group 3 (MenC-Primed): MenACYW Conjugate Vaccine vs Group 4 (MenC-Primed): Nimenrix®; Serogroup A; Test type: Other; GMT Ratio = 0.496, 95% CI 2-sided [0.367 to 0.672]
Statistical Analysis 2: Comparison: Group 3 (MenC-Primed): MenACYW Conjugate Vaccine vs Group 4 (MenC-Primed): Nimenrix®; Serogroup C; Test type: Other; GMT Ratio = 1.34, 95% CI 2-sided [0.814 to 2.19]
Statistical Analysis 3: Comparison: Group 3 (MenC-Primed): MenACYW Conjugate Vaccine vs Group 4 (MenC-Primed): Nimenrix®; Serogroup Y; Test type: Other; GMT Ratio = 1.53, 95% CI 2-sided [1.15 to 2.04]
Statistical Analysis 4: Comparison: Group 3 (MenC-Primed): MenACYW Conjugate Vaccine vs Group 4 (MenC-Primed): Nimenrix®; Serogroup W; Test type: Other; GMT Ratio = 1.29, 95% CI 2-sided [0.944 to 1.75]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to 30 days after vaccination. Solicited Reactions (SRs) data were collected within 7 days after vaccination. Serious adverse events (SAEs) data were collected throughout the study (up to 30 days after vaccination).
Description: Analysis was performed on Safety Analysis Set. A SR was an AE that was prelisted (i.e.solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e.solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine | Group 2 (Meningococcal Vaccine-Naive): Nimenrix® | Group 3 (MenC-Primed): MenACYW Conjugate Vaccine | Group 4 (MenC-Primed): Nimenrix®
All-Cause Mortality (participants affected / at risk) | 0/303 | 0/306 | 0/203 | 0/102
Serious Adverse Events (participants affected / at risk) | 2/303 | 1/306 | 2/203 | 2/102
Other Adverse Events (participants affected / at risk) | 261/303 | 266/306 | 151/203 | 65/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine (N=303) | Group 2 (Meningococcal Vaccine-Naive): Nimenrix® (N=306) | Group 3 (MenC-Primed): MenACYW Conjugate Vaccine (N=203) | Group 4 (MenC-Primed): Nimenrix® (N=102)
Haemolytic Uraemic Syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Malrotation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Campylobacter Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Escherichia Coli (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Immunoglobulin A Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1(Meningococcal Vaccine-Naive):MenACYW Conjugate Vaccine (N=303) | Group 2 (Meningococcal Vaccine-Naive): Nimenrix® (N=306) | Group 3 (MenC-Primed): MenACYW Conjugate Vaccine (N=203) | Group 4 (MenC-Primed): Nimenrix® (N=102)
Diarrhoea (Gastrointestinal disorders) | 23 (23) | 16 (16) | 8 (8) | 4 (4)
Teething (Gastrointestinal disorders) | 16 (18) | 13 (19) | 12 (15) | 6 (7)
Vomiting (Gastrointestinal disorders) | 23 (24) | 13 (13) | 21 (21) | 8 (8)
Crying (General disorders) | 106 (109) | 111 (112) | 48 (48) | 23 (23)
Injection Site Erythema (General disorders) | 122 (123) | 116 (116) | 52 (52) | 21 (21)
Injection Site Pain (General disorders) | 122 (122) | 113 (113) | 55 (55) | 20 (21)
Injection Site Swelling (General disorders) | 63 (63) | 52 (52) | 35 (35) | 9 (9)
Pyrexia (General disorders) | 40 (42) | 48 (48) | 29 (29) | 14 (15)
Bronchitis (Infections and infestations) | 3 (4) | 2 (2) | 11 (11) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (19) | 18 (18) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 21 (22) | 25 (27) | 5 (5) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 49 (55) | 39 (43) | 14 (14) | 7 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 91 (93) | 94 (94) | 56 (56) | 28 (28)
Somnolence (Nervous system disorders) | 64 (64) | 55 (55) | 51 (51) | 19 (19)
Irritability (Psychiatric disorders) | 144 (145) | 127 (128) | 76 (76) | 36 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 13 (16) | 13 (13) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT02955797/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT02955797/SAP_001.pdf